CLINICAL TRIAL: NCT04721444
Title: Optimising Cancer Therapy And Identifying Causes of Pneumonitis USing Artificial Intelligence
Brief Title: Optimising Cancer Therapy And Identifying Causes of Pneumonitis USing Artificial Intelligence (COVID-19)
Acronym: OCTAPUS-AI
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 5293
Record Dates: First submitted 2020-11-06; First posted 2021-01-22 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Lung Cancer; Covid19; Pneumonitis
MeSH Terms: conditions — Lung Neoplasms; COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Arm A - Cohort A1: Training set: Pneumonitis in the context of IO therapy and negative for infectious pneumonia (including COVID-19)
  Interventions: Diagnostic Test: Machine Learning Classification of parenchymal lung change cause
- Arms A and B - Cohort B1: Training set B1: IO and RT naive and pneumonia (without COVID-19)
  Interventions: Diagnostic Test: Machine Learning Classification of parenchymal lung change cause
- Arms A and B - Cohort B2: Training set B2: IO and RT naive and confirmed COVID-19 positive with pneumonia
  Interventions: Diagnostic Test: Machine Learning Classification of parenchymal lung change cause
- Arm B - Cohort A2: Training set: Pneumonitis in the context of thoracic RT and negative for infectious pneumonia (including COVID-19)
  Interventions: Diagnostic Test: Machine Learning Classification of parenchymal lung change cause
- Arm A - Test Cohort (Cohort C1): Test set C1: Patients on IO and with possible toxicity versus COVID-19 or other infective pneumonitis
  Interventions: Diagnostic Test: Machine Learning Classification of parenchymal lung change cause
- Arm B - Test Cohort (Cohort C2): Test set C2: Patients with pneumonitis in context of thoracic RT with possible toxicity versus COVID-19 or other infective pneumonitis.
  Interventions: Diagnostic Test: Machine Learning Classification of parenchymal lung change cause
- Arm C: Patients with radiotherapy planning CT scans and post-treatment surveillance CT scans at 3, 6 and 12-months post treatment
  Interventions: Diagnostic Test: Machine Learning Classification of recurrence and non-recurrence

INTERVENTIONS:
Diagnostic Test: Machine Learning Classification of parenchymal lung change cause — Arms A & B: Radiomics and deep-learning approaches will be used on patient's imaging to develop a feature vector that can distinguish parenchymal lung changes, e.g. infection from drug-toxicity.
  Groups: Arm A - Cohort A1; Arm A - Test Cohort (Cohort C1); Arm B - Cohort A2; Arm B - Test Cohort (Cohort C2); Arms A and B - Cohort B1; Arms A and B - Cohort B2
Diagnostic Test: Machine Learning Classification of recurrence and non-recurrence — Arm C: Radiomics and deep-learning approaches will be used on patient's imaging to develop a risk-signature for recurrence of malignancy following radical treatment
  Groups: Arm C

SUMMARY:
Distinguishing changes on patients that have received thoracic radiotherapy and patients that are currently receiving or have recently received IO and presenting lung changes which will be identified using AI.

ELIGIBILITY:
Arms A & B:

Inclusion Criteria:

Cohort A1 (from Arm A) - Immunotherapy (IO) pneumonitis cases: patients currently on or having received ICI IO in the last 3 months of presentation with:

• New radiological lung changes on CT/CXR (confirmed on report) of a severity and distribution consistent with IO pneumonitis. These changes should be of severity and distribution that are not incompatible with viral or lower respiratory tract infection.

AND Must not have had RT involving the thorax (unless this was breast/chest wall RT more than 5 years ago, which is permissible) AND

* Where there is documented clinical concern for infection, have undergone one or more laboratory investigations for viral or lower respiratory tract infection including, but not limited to Nasopharyngeal aspirate or swab for respiratory virus by PCR; Sputum sample or bronchial washings MCS with no organism(s) consistent with lower respiratory tract infection, cytology or beta-glucan/galactomannan for PCP or fungal infection; broncho-alveolar lavage for markers of infection such as MCS, PCR, fungal culture, beta-glucan/galactomannan for PCP or evidence of lower respiratory tract infection (including invasive fungal infection) by cytology, none of which were considered positive for infection by the clinical team.
* Where empirical antibiotics were prescribed, patients must either have had a negative BAL infection screen or may be included at the discretion of the local site PI and local radiologist with lung interest or two members of the trial management group, one of whom must be a radiologist with lung interest or respiratory physician or oncologist with suitable experience of thoracic CT imaging, after after review of the case-notes.
* Prophylactic co-trimoxazole prescribed in the context of high-dose steroid therapy is permitted.

Cohort A2 (from Arm B) - Radiotherapy (RT) pneumonits cases: Patients that have completed a course of RT involving the thorax (e.g. lung, breast, oesophageal RT) in the last 12 months prior to presentation, that have not received immunotherapy, with:.

• New radiological lung changes on CT/CXR (confirmed on report) of a severity and distribution consistent with radiation pneumonitis or early fibrosis (should not include established fibrosis). These changes should be of severity and distribution that are not incompatible with viral or lower respiratory tract infection.

AND

* Where there is documented clinical concern for infection, have undergone one or more laboratory investigations for viral or lower respiratory tract infection including, but not limited to Nasopharyngeal aspirate or swab for respiratory virus by PCR; Sputum sample or bronchial washings MCS with no organism(s) consistent with lower respiratory tract infection, cytology or beta-glucan/galactomannan for PCP or fungal infection; broncho-alveolar lavage (BAL) for markers of infection such as MCS, PCR, fungal culture, beta-glucan/galactomannan for Pneumocystis Pneumonia (PCP) or evidence of lower respiratory tract infection (including invasive fungal infection) by cytology, none of which were considered positive for infection by the clinical team. Where empirical antibiotics were prescribed, patients must either have had a negative BAL infection screen or may be included at the discretion of the local site PI and local radiologist with lung interest or two members of the trial management group, one of whom must be a radiologist with lung interest or respiratory physician or oncologist with suitable experience of thoracic CT imaging, after review of the case-notes.
* Prophylactic co-trimoxazole prescribed in the context of high-dose steroid therapy is permitted.

B1 (Utilised in Arms A & B) Non-COVID-19 infective cases:

* New radiological lung changes on CT/CXR (confirmed on report) of a severity and distribution consistent with lower respiratory tract infection but compatible with the grade and nature of pneumonitis seen with IO or RT
* AND
* Laboratory findings that fulfil one or more of the following criteria of infection: Nasopharyngeal aspirate or swab positive for a respiratory virus by PCR; Sputum sample or bronchial washings positive MCS for an organism(s) consistent with lower respiratory tract infection, cytology or beta-glucan/galactomannan positive for PCP or fungal infection, positive urine legionella/pneumococcal antigen screen, positive serology for mycoplasma pneumonia; broncho-alveolar lavage for markers of infection (MCS, PCR, fungal culture, beta-glucan/galactomannan for PCP or other evidence of lower respiratory tract infection (including invasive fungal infection) by cytology. Where no such laboratory findings were positive but the patient improved with anti-microbial therapy, such cases may be included at the discretion of the local site PI and local radiologist with lung interest or two members of the trial management group two members of the trial management group, one of whom must be a radiologist with a lung interest or respiratory physician or oncologist with suitable experience of thoracic CT imaging, after review of the case-notes and imaging.
* Not previously treated with immunotherapy OR
* Must not have had RT involving the thorax (unless this was breast/chest wall RT more than 5 years ago, which is permissible)
* First assessed prior to 1st January 2020 (and therefore not attributable to COVID-19)

B2 (Utilised in Arms A & B) COVID-19 cases:

• Laboratory findings that fulfil one or more of the following criteria of COVID-19 infection: positive COVID-19 PCR test and/or antigen test or other suitable assay that indicates current infection or previous exposure (including serology tests) as determined by the trial management group (TMG).

AND

* New radiological lung changes on CT/CXR (confirmed on report) of a severity and distribution consistent with COVID-19. These changes should be of severity and distribution that is not incompatible with the grade of pneumonitis seen with IO or RT
* Not previously treated with immunotherapy OR
* Must not have had RT involving the thorax (unless this was breast/chest wall RT more than 5 years ago, which is permissible)
* Assessed after 1st January 2020 (and therefore contemporaneous with COVID-19)

Exclusion Criteria:

• Patients with documented past medical history of congestive cardiac failure or other cause for interstitial lung disease

Arm C:

Inclusion Criteria:

* Adult patients (aged 18 or over) treated with radical thoracic RT (conventional fractionated RT +/- chemotherapy or SBRT) for NSCLC
* RT planning scan imaging and labelled structure set data available from participating centre
* Minimum 2 years of post-RT follow-up data including clinical or histological confirmation in the case of recurrence and whether the patient is alive as available from primary care or hospital records.
* Patients with post-treatment surveillance CT imaging (minimum of first scan post-treatment and where available +/- further scans within 2 years post-RT, e.g. at 3/6/12 months post-treatment).

Exclusion Criteria:

* Any patient that does not have a primary lung mass e.g. Tx disease
* Any patient being treated for recurrence of a previously treated lung cancer
* Any patient that did not have radical RT e.g. patients that had high dose palliative RT
* Any patient that does not have imaging that meets technical requirements within the imaging processing and analysis manual

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Arms A and B: Adult patients with pneumonitis that have previously been treated with thoracic radiotherapy or immunotherapy Arm C: Adult patients that have received radical radiotherapy for NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 1211 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Development of a Machine Learning model to distinguish parenchymal lung changes | 3 years
  The development and validation of an ML/radiomic classifier to distinguish between Infective/COVID-19 pneumonia and cancer therapy induced lung changes
Development of a Machine Learning model to predict recurrence risk after radical radiotherapy for non-small cell lung cancer | 3 years
  to develop a prognostic AI/radiomic signature for NSCLC recurrence after radical RT (Conventional fractionated RT +/- chemotherapy or stereotactic body RT (SBRT)) to stratify appropriate surveillance and onward care, thus minimising unnecessary hospital visits and resource use.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lee, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Guys and St. Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Royal Marsden NHS Foundation Trust, London